CLINICAL TRIAL: NCT05763654
Title: Multicenter, Long-term, Single-arm and Observational PMCF Study on the Safety of Linovera Emulsion for the Prevention of Stage 1 Pressure Ulcers, Vascular and Diabetic Foot Ulcers (PRELINEM)
Brief Title: PMCF Study on the Safety of Linovera Emulsion for the Prevention of Cat-1 Pressure Ulcers, Vascular and DFU
Acronym: PRELINEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: BA-G-H-2201
Record Dates: First submitted 2022-11-25; First posted 2023-03-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Linovera emulsion: No intervention. Routine clinical practice.
  Interventions: Device: Linovera emulsion

INTERVENTIONS:
Device: Linovera emulsion — Apply Linovera emulsion in clinical routine

SUMMARY:
To assess the safety of Linovera® Emulsion in the prevention of Grade I Pressure ulcers, Vascular and Diabetic Foot Ulcers.

To assess the performance of Linovera® Emulsion for the prevention of stage 1 Pressure Ulcers, Vascular and Diabetic Foot Ulcers.

DETAILED DESCRIPTION:
Diverse parameters are to be used to assess the safety and efficacy of Linovera® Emulsion for the prevention of stage 1 pressure ulcer, vascular and diabetic foot ulcers.

This study is designed to implement an action within the framework of a proactive Post Market Clinical Follow up (PMCF) activity as a part of our Post Market Surveillance (PMS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed informed consent
* Patients with the possibility to participate during up 6 month follow-up.
* At least one of these criteria:
* Patients with medium, high or very high risk of amputation due to a vascular or diabetic foot illness.
* Patients with medium, high or very high risk of developing a pressure ulcer due to any neuropathic foot pathology
* Patients with medium, high or very high risk of developing a pressure ulcer following Braden Scale.

Exclusion Criteria:

* Age < 18 years
* Known allergies and/or hypersensitivity to any component of Linovera® Emulsion.
* Any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to give informed consent and comply with the study procedures.
* Patients in the terminal stage or receiving chemotherapy.
* Patients with more than 3 active pressure ulcers.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Already described in Inclusion and Exclusion criteria
Sampling Method: Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 1 month
  Number of adverse events

SECONDARY OUTCOMES:
Number of participant developing stage 1 Pressure Ulcers, Vascular and Diabetic Foot Ulcers | 1 month
  Number of participants developing stage 1 Pressure Ulcers, Vascular and Diabetic Foot Ulcers

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Alvaro Cunqueiro, Vigo, Spain

IPD SHARING:
Plan to Share IPD: Undecided